CLINICAL TRIAL: NCT06433050
Title: Sodium Glucose Co-transporter (SGLT) Inhibitors in Nonobstructive Hypertrophic Cardiomyopathy
Acronym: SOTA-CROSS HCM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sharlene Day, Associate Professor of Cardiovascular Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 855065; R61HL164376 (NIH)
Record Dates: First submitted 2024-05-13; First posted 2024-05-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hypertrophic Cardiomyopathy Without Obstruction
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo first phase, Sotagliflozin second phase (Placebo Comparator): Matching placebo once daily will be administered in the first phase, Sotagliflozin 400 mg once daily will be administered in the second phase
  Interventions: Drug: Sotagliflozin
- Sotagliflozin first phase, Placebo second phase (Active Comparator): Sotagliflozin 400 mg once daily will be administered in the first phase, matching placebo once daily will be administered in the second phase
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin or placebo will be administered to each participant in a cross over study design. Each participant will receive active drug and placebo with randomization of the order in which they receive them.
  Other Names: Inpefa

SUMMARY:
The goal of this clinical trial is to learn if sotagliflozin, a dual SGLT1 and SGLT2 inhibitor, works to treat symptomatic, nonobstructive hypertrophic cardiomyopathy (noHCM) in adult patients. It will also learn about the safety of sotagliflozin in this patient population. The main questions it aims to answer are:

1. Will sotagliflozin be well tolerated in patients with nonobstructive HCM?
2. Will sotaglifozin improve exercise capacity, diastolic dysfunction and/or physical functioning in patients with nonobstructive HCM?
3. Will sotagliflozin improve circulating markers of cardiac metabolism in patients with nonobstructive HCM?

Researchers will compare sotagliflozin to a placebo (a look-alike substance that contains no drug) to see if sotagliflozin is effective at treating hypertrophic cardiomyopathy (HCM).

Participants will:

Take sotagliflozin or a placebo every day for 12 weeks. They will then cross-over (or switch) to taking placebo or sotagliflozin (whichever one they did not take initially) for an additional 12 weeks.

Visit the clinic once every 4-12 weeks for checkups, surveys, and tests including a stress test and echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years, both sexes
2. Provision of signed and dated informed consent form
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Ability to take oral medication and be willing to adhere to the study intervention.
5. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 2 weeks after the end of administration of study drug.
6. Diagnosis of HCM with NYHA Class II-III functional class or New York Heart Association (NYHA) Class I with peak VO2 < 90% on cardiopulmonary exercise stress testing performed at Visit 1.
7. Left ventricular outflow tract gradient < 50 mmHg at rest, with valsalva, and with exercise.

7. Left ventricular ejection fraction > 50% by echocardiogram or cardiac MRI based on the most recent assessment in the past year prior to screening and confirmed during Visit 1 echocardiogram.

8. Stable medical therapy for at least 1 month prior to study enrollment.

Exclusion Criteria:

1. Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrollment or previous intolerance of an SGLT2 inhibitor
2. Type 1 diabetes mellitus
3. Age <18 years old
4. Pregnant or lactating women: Women of childbearing potential will undergo a urine pregnancy test during the screening visit.
5. Uncontrolled atrial fibrillation, as defined by a resting heart rate > 100 beats per minute at the time of the baseline assessment
6. Paroxysmal atrial fibrillation (Afib) or flutter with plans to attempt to restore sinus rhythm (with drug therapy, ablation, or DC cardioversion) during the study period.
7. Unable to attain a respiratory exchange ratio of at least 1.05 on cardiopulmonary exercise test (CPET) on the day of screening.
8. Septal reduction therapy within the previous 3 months.
9. Implantable cardio-defibrillator (ICD) implantation planned during the study period.
10. Implantation of a cardiac resynchronization therapy (CRT) device within 12 weeks prior to enrollment or intent to implant a CRT device during the study period
11. Hemoglobin < 10 g/dL
12. Estimated glomerular filtration rate (eGFR) < 25 mL/min/1.73m^2, or unstable or rapidly progressing renal disease at the time of randomization
13. Subject inability/unwillingness to exercise
14. Greater than moderate left sided valvular disease (mitral regurgitation, aortic stenosis, aortic regurgitation), moderate or greater mitral stenosis, or severe right-sided valvular disease based on baseline echo at the time of enrollment
15. Current angina due to clinically significant epicardial coronary disease, as per investigator judgment
16. Acute coronary syndrome or coronary intervention within the past 2 months
17. Primary pulmonary artery hypertension (WHO Group 1 Pulmonary Arterial Hypertension)
18. Clinically significant lung disease as defined by: Chronic Obstructive Pulmonary Disease meeting Stage III or greater GOLD criteria (FEV1<50% predicted), treatment with oral steroids within the past 6 months for an exacerbation of obstructive lung disease, or current use of supplemental oxygen aside from nocturnal oxygen for the treatment of obstructive sleep apnea.
19. Clinically-significant ischemia, as per investigator's judgement, on stress testing without either (1) subsequent revascularization, (2) an angiogram demonstrating the absence of clinically significant epicardial coronary artery disease, as per investigator judgment; (3) a follow-up 'negative' stress test, particularly when using a more specific technique (i.e., a negative perfusion imaging test following a 'positive' ECG stress test)
20. Symptomatic bradycardia or second- or third-degree heart block, in the absence of a pacemaker
21. Significant liver disease impacting synthetic function or volume control (ALT/AST > 3x ULN, Albumin < 3.0 g/dL)
22. Severe right ventricular dysfunction on baseline echocardiogram
23. Orthostatic blood pressure response to the transition from supine to standing (>20 mmHg reduction in systolic blood pressure 2-3 minutes after standing)
24. Active participation in another study that utilizes an investigational agent (observational studies/registries allowed)
25. Any condition that, in the opinion of the investigator, will interfere with the completion of the study. This may include comorbid or psychiatric conditions that may impede successful completion of the protocol, or logistical concerns (e.g. inability to travel to the exercise unit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | Through study completion, 28 weeks
  Adverse event reporting
Intracavitary obstruction | Through study completion, 28 weeks
  Intracavitary left ventricular pressure gradient in mmHg
Cardiac rhythm | Through study completion, 28 weeks
  New occurrence of cardiac arrhythmia measured by ambulatory monitoring
Maximal exercise capacity | Through study completion, 28 weeks
  Peak oxygen consumption in mL/min
Submaximal exercise capacity | Through study completion, 28 weeks
  Stroke volume augmentation at exercise steady state in mL/min

SECONDARY OUTCOMES:
Systolic function | Through study completion, 28 weeks
  Left ventricular ejection fraction in % measured by echocardiography
Contractility | Through study completion, 28 weeks
  Global longitudinal strain in % measured by echocardiography
Diastolic function | Through study completion, 28 weeks
  E/E' ratio measured by echocardiography
Left ventricular hypertrophy | Through study completion, 28 weeks
  Maximal left ventricular wall thickness in mm by echocardiography
Symptom scores | Through study completion, 28 weeks
  Kansas City Living with Heart Failure (KCCQ) Clinical Summary Score, scale 0-100 with lower scores being worse
Symptom scores and quality of life | Through study completion, 28 weeks
  Kansas City Living with Heart Failure (KCCQ) Overall Summary Score, score 0-100 with lower scores being worse
Biomarkers | Through study completion, 28 weeks
  Serum levels of N-terminal-proBNP
Circulating metabolites | Through study completion, 28 weeks
  Concentration of serum metabolites
Measurement of periods of activity and rest | Through study completion, 28 weeks
  Daily step counts by actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Sharlene Day, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers